CLINICAL TRIAL: NCT02626247
Title: Effect of Lipidic Nutrients on Memory and Well Being in Healthy Aging Adults
Acronym: NUTRIMEMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutrimemo Consortium (Other)
Collaborators: University of Bordeaux (Other); Unither Pharmaceuticals, France (Industry); Company Groupe St Hubert France (Unknown); VAB Nutrition France (Unknown); ITERG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2015-08-28; First posted 2015-12-10 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: elderly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin A + Long chain PUFA (Active Comparator): The test product is a food supplement containing Vitamin A + Long chain Poly Unsaturated Fatty Acids (PUFA). It is presented as a hard shell capsule containing lipophylic nutrients.
  Interventions: Dietary Supplement: Vitamin A +Long chain PUFA
- Placebo (Placebo Comparator): The placebo is a capsule with same appearance and organoleptic properties as the active product, containing no active component.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin A +Long chain PUFA — 3 capsules per day, two capsules at breakfast and one capsule at lunch, with a glass of water.
  Arms: Vitamin A + Long chain PUFA
Other: Placebo — 3 capsules per day, two capsules at breakfast and one capsule at lunch, with a glass of water.
  Arms: Placebo

SUMMARY:
Nutrimemo aims to study the effect of a daily consumption of a mix of vitamin A and long chain n-3 Polyunsaturated Fatty Acids (PUFA) on the evolution of cognitive functions in healthy elderly subjects. The study is a randomized, double bind, parallel-groups (2 arms) placebo-controlled design.

DETAILED DESCRIPTION:
This project aims to investigate the effects of 12 months supplementation with a mix of Vitamin A + Long chain n-3 PUFA vs placebo to consume daily on human cognitive functions. Food supplement and placebo will be provided as capsules matched for appearance.

The study will be conducted as a randomized, double-blind, parallel-groups (2 arms) placebo-controlled. Two groups, each of 180 volunteers, are recruited. One group of volunteers will consume the Vitamin A + Long chain n-3 PUFA mix while the other one will consume the placebo product.

Each volunteer will be seen for 5 visits at the investigational site. Baseline and the last follow-up visit will include cognitive assessment with the CANTAB battery. CANTAB tests will cover several aspects of memory: visio-spatial learning and episodic memory, visio-spatial working memory, frontal executive functions, but also word-based semantic memory.

Moreover, psychological and mood components will be evaluated (mnesic complaint, depression, fatigue). Physical activity will also be recorded. Finally, biological parameters will be assessed (lipid profile, glycemia, CRP, thyroid stimulating hormone, transthyretin, plasma level of vitamin A and D as well as retinol binding protein and lipidic profile).

ELIGIBILITY:
Inclusion Criteria:

* Independent subjects
* Living at home non diagnosed as Alzheimer
* Body Mass Index (BMI) 20-30 kg/m2 (limits included);
* 26 < MMSE score ≤ 29
* Logical memory subtest of the Wechsler Memory Scale (16-69 years battery) - sub-scores complying with the following:

  * Immediate recall score < 29;
  * Delayed recall score < 16;

Exclusion Criteria:

* Evidence of actual major depressive disorder according to the module A of the Mini International Neuropsychiatric Interview (MINI);
* Subject consuming food supplements likely to have an effect on memory or within less than 6 months;
* Subject consuming high level of Vitamin A and/or Long chain n-3 PUFA evaluated by a food frequency questionnaire,
* Restrictive or unbalanced diet (hypocaloric, vegetarian, vegan, …) self-declared at V0;
* Alcohol consumption > 4 glasses/day
* Diabetes;
* Cardiovascular disease diagnosed within less than 2 years, with the following exceptions: subjects with controlled (medicated) high blood pressure and/ or controlled (medicated) can be included;
* Unbalanced thyroid disease;
* Anti-depressant treatment stopped since less than 3 months or still ongoing;
* Personal history of schizophrenia or other psychiatric disorders;
* Ongoing neuroleptic treatment;
* Uncorrected visual or auditory dysfunction (according to the volunteer's self-declaration);
* Life threatening pathology (such as cancer) in remission for less than 1 year or still ongoing;
* General anesthesia in the last 6 months or planned in the next 6 months;
* Documented food allergy(ies), namely to one of the components of the study product;
* Psychological or linguistic incapability to sign the informed consent.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline of the episodic memory measured by CANTAB - Paired Associate Learning test (PAL) | 52 weeks

SECONDARY OUTCOMES:
Change From Baseline of the working memory measured by CANTAB - Spatial Span test (SSP) | 52 weeks
Change From Baseline of the executive function and spatial planning measured by CANTAB - One tone Touch Stockings of cambridge " (OTS) | 52 weeks
McNair scale | 52 weeks
  The McNair and Kahn scale is a subjective scale used to evaluate the memory complaints in front of everyday conditions.
Change from baseline of the Verbal fluency measured by Isaac verbal fluency test | 52 weeks
  Isaac verbal fluency test is a test for semantic memory and verbal fluency. The test consists to ask the patient to name in 15 seconds the most possible words around 4 semantic categories: colors, animals, fruits, cities (10 responses by category and score/40).
Montgomery et Asberg Depression Scale | 52 weeks
COVI anxiety Scale | 52 weeks
Change From Baseline in Mini-Mental State Examination (MMSE) | 52 weeks
  The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline.
Multidimensional Fatigue Inventory (MFI-20) | 52 weeks
SF36 (Medical Outcome Study, Short-Form 36) | 52 weeks
blood lipidic profile | 52 weeks
  Cholesterol g/L and Triglycerides g/L
Glycemia | 52 weeks
  g/L
blood hight sensitive C reactive Protein (CRP) | 52 weeks
  mg/L
blood Retinol | 52 weeks
  µM/L
Blood retinol binding protein (RBP) | 52 weeks
  mg/L
Blood transtyretin | 52 weeks
  g/L
salivary cortisol | 52 weeks
  nmol/L
blood free Thyroxine | 52 weeks
  g/L
Blood triiodothyronine | 52 weeks
  pg/MmL
blood Vitamin D 25 OH | 52 weeks
  nmol/L
Fatty acid profile in erythrocyte membranes | 52 weeks
  % of total fatty acids
Nuclear receptor mRNA expression in mononuclear cells | 52 weeks
  relative expression
blood Inflammatory markers | 52 weeks
  g/L
plasma beta amyloide | 52 weeks
  pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Véronique PALLET, Professor, Study Director — Laboratoire NutriNeuro INRA-Université de Bordeaux
Locations (1):
- Universitary Hospital Center - USR 3413 SANPSY, Bordeaux, France

REFERENCES:
- See also: website of the laboratory of Nutrition and integrative neurobiology (NutriNeuro) — http://www6.bordeaux-aquitaine.inra.fr/nutrineuro